CLINICAL TRIAL: NCT01839123
Title: Prosthetic Socket System: Pilot Assessment
Brief Title: Evaluation of Limb Health Associated With a Prosthetic Vacuum Socket System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ohio Willow Wood (Industry)
Collaborators: Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: VA-2012-Aim1; VA118-12-C-0038 (Other Grant/Funding Number: Veterans Affairs Innovation Initiative)
Record Dates: First submitted 2013-04-19; First posted 2013-04-24 (Estimated); Last update posted 2013-07-01 (Estimated); Status verified 2013-06

CONDITIONS: Lower Limb Amputation
Keywords: Amputee

ARMS (2):
- Non-Vacuum Socket (Active Comparator): Prosthetic suction or pin socket
  Interventions: Device: Prosthetic Suction or Pin Socket
- Vacuum Socket (Experimental): Prosthetic LimbLogic vacuum socket
  Interventions: Device: Prosthetic LimbLogic Vacuum Socket

INTERVENTIONS:
Device: Prosthetic Suction or Pin Socket — Conventional prosthetic socket utilizing non-vacuum suspension to secure the residual limb to the prosthesis. Non-vacuum suspension includes pin/lock suspension and suction suspension.
  Other Names: Pin and Lock Suspension; Pin Socket; Suction Suspension; Suction Socket
  Arms: Non-Vacuum Socket
Device: Prosthetic LimbLogic Vacuum Socket — Prosthetic socket that incorporates conventional vacuum suspension using the commercially available LimbLogic vacuum pump
  Arms: Vacuum Socket

SUMMARY:
The purpose of the study is to evaluate residual limb circulation and skin health associated with the use of a prosthetic vacuum socket. A conventional non-vacuum prosthetic socket will be compared to a vacuum prosthetic socket.

DETAILED DESCRIPTION:
The prosthetic suspension plays a pivotal role in an amputee's comfort. It can also significantly impact an amputee's limb health. If the prosthesis is not held securely to the amputee's limb, relative movement between the limb and prosthetic interface can cause bruising, skin irritation and skin breakdown. These poor outcomes are uncomfortable and can lead to much more serious health conditions. A positive solution to creating secure and comfortable suspension is the use of a vacuum suspension socket. The vacuum pressure assists in preventing movement in the socket. The clinical benefits associated with vacuum suspension include volume retention, increased proprioception, secure suspension, and frequently reported observations of wound healing. However, the long term effects of vacuum suspension on circulation remain undetermined or undocumented.

This study examines a vacuum suspension system on the health of the residual limb (amputated limb). A vacuum socket creates a vacuum between the rigid prosthetic socket and prosthetic liner which is sealed to the socket. Therefore, vacuum is not directly applied to the skin of the residual limb.

ELIGIBILITY:
Inclusion Criteria:

* Consenting Adult
* Unilateral lower extremity amputee
* Currently using a liner with prosthesis
* Uses a prosthesis to ambulate
* Ability to read, write and understand English
* Available during regular business hours for appointments

Exclusion Criteria:

* Impaired contra lateral leg
* Uses vacuum suspension with their current prosthesis
* Diagnosis of renal failure
* Smoker

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2013-04; Primary Completion 2014-09 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Transcutaneous partial pressure of oxygen (tcpO2 level) at 16 wks | 16 weeks
  Change from baseline in Transcutaneous partial pressure of oxygen (tcpO2 level) at 16 wks

SECONDARY OUTCOMES:
Transcutaneous partial pressure of oxygen (tcpO2 level) at 8 wks | 8 weeks
  Change from baseline in Transcutaneous partial pressure of oxygen (tcpO2 level) at 8 wks
Hyperspectral Imaging Tissue Oxygen Saturation (StO2%) at 8wks | 8 weeks
  Change from baseline in Hyperspectral Imaging StO2% at 8wks
Hyperspectral Imaging StO2% at 16wks | 16 weeks
  change from baseline in Hyperspectral Imaging StO2% at 16wks
Laser speckle flowmetry tissue perfusion values at 8wks | 8 weeks
  Change from baseline in Laser speckle flowmetry tissue perfusion values at 8wks
Laser speckle flowmetry tissue perfusion values at 16wks | 16 weeks
  Change from baseline in Laser speckle flowmetry tissue perfusion values at 16wks
Laser Doppler flowmetry tissue perfusion values at 8wks | 8 weeks
  Change from baseline in Laser Doppler flowmetry tissue perfusion values at 8wks
Laser Doppler flowmetry tissue perfusion values at 16wks | 16 weeks
  Change from baseline in Laser Doppler flowmetry tissue perfusion values at 16wks

OTHER OUTCOMES:
Skin temperature values at 8wk | 8 weeks
Prosthesis evaluation questionnaire (PEQ) | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gayle Gordillo, MD, Principal Investigator — Ohio State University
Locations (2):
- United States (2):
  - The Ohio State University Davis Heart and Lung Research Institute, Columbus, Ohio
  - The Ohio Willow Wood Company, Mount Sterling, Ohio

REFERENCES:
- [Derived] Rink C, Wernke MM, Powell HM, Gynawali S, Schroeder RM, Kim JY, Denune JA, Gordillo GM, Colvin JM, Sen CK. Elevated vacuum suspension preserves residual-limb skin health in people with lower-limb amputation: Randomized clinical trial. J Rehabil Res Dev. 2016;53(6):1121-1132. doi: 10.1682/JRRD.2015.07.0145. PMID 28355039